CLINICAL TRIAL: NCT03299348
Title: Testing Psychological Mechanisms to Promote Physical Activity in Adults
Brief Title: AgingPLUS: Promoting Physical Activity in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: Johns Hopkins University (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Manfred Diehl, PhD, Professor, Colorado State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 3437; 5R01AG051723-05 (NIH)
Record Dates: First submitted 2017-09-23; First posted 2017-10-03 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Physical Activity
Keywords: Psychological Mechanisms; Social-Cognitive Mechanisms
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study has an active treatment group and an active control group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Study participants, group leaders, and outcomes assessors will not know the study objectives or hypotheses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Treatment Group (Experimental): This group will get the AgingPLUS intervention program which addresses negative views on aging, low internal control beliefs, and deficient goal planning skills.
  Interventions: Behavioral: AgingPLUS
- Active Control Group (Placebo Comparator): This group will get a generic health education program, called the "10 Keys to Healthy Aging". The control program will control for the effect of social contact and will not address the intervention targets of the active treatment group. The health education program will only provide information related to some of the most important health conditions, such as cardiovascular disease, cancer, type 2 diabetes, and clinical depression, and how these conditions can be managed.
  Interventions: Behavioral: Active Control Group

INTERVENTIONS:
Behavioral: AgingPLUS — The program consists of 2-hour meetings for a total of 4 weeks (total of 8 hours) and discusses (a) how negative views on aging and negative age stereotypes undermine adults' health-promoting behaviors; (b) how adults can take control of their own aging; and (c) how personal goals can be achieved through more effective goal planning and action plans.
  Arms: Active Treatment Group
Behavioral: Active Control Group — The program consists of 2-hour meetings for a total of 4 weeks (total of 8 hours) and discusses (a) four major health conditions that affect the lives of many middle-aged and older adults (e.g., cardiovascular disease, cancer, type 2 diabetes; clinical depression); and (b) how these conditions can be managed successfully.
  Arms: Active Control Group

SUMMARY:
This study examines the efficacy of a psycho-educational intervention program, AgingPLUS, with regard to increasing middle-aged and older adults' engagement in physical activity.

DETAILED DESCRIPTION:
AgingPLUS is a multi-component intervention program that addresses negative views of aging (NVOA), low internal control beliefs, and deficient goal planning as a risk cluster that keeps adults from engaging in health-promoting behavior. The program focuses on engagement in physical activity (PA) as the health behavior of choice. Engagement in PA is widely recognized as the best non-pharmacological, non-invasive, and cost-effective method of health promotion. Yet, only 20% of the adult population meets the recommended PA guidelines. This suggests that messages about the benefits of PA alone are not effective. Rather, it is essential to address the social-cognitive and motiva-tional mechanisms that prevent adults from adopting and maintaining a regular PA regimen. NVOA, low internal control beliefs, and deficient goal planning represent such a cluster of social-cognitive and motivational mechanisms.

Given this background, the specific aims and hypotheses of the proposed research are:

Aim 1: To conduct a randomized controlled trial examining the efficacy of the AgingPLUS program.

Aim 2: To test a conceptual model of the mechanisms underlying the intervention effects.

Aim 3: To conduct a 6-month follow-up to examine the longer-term effects of AgingPLUS.

Upon completion of this project, we expect to have successfully established evidence for the efficacy of the AgingPLUS program (Stage II of the NIH Stage Mode). The long-term goal is to develop AgingPLUS into a full-fledged evidence-based program that can be implemented in community settings (e.g., senior centers), and can serve as a fairly brief and cost-effective public health tool to promote healthy and successful aging.

ELIGIBILITY:
Inclusion Criteria:

* Adults who engage in less than 60 minutes of PA per week and who intend starting a physical exercise program.
* English speaking.
* Willingness to be randomized to one of two programs.
* Willingness to take part in the physical fitness tests and wear an accelerometer.
* Willingness to commit to follow-up testing (i.e., not moving out of the area during the study period).
* Physician clearance to take part in a submaximal exercise test and to begin an exercise program.

Exclusion Criteria:

* Signs of cognitive decline (defined as more than 4 errors on the Short Portable Mental Status Questionnaire).
* Severe vision and/or hearing loss (obtained by self-report).
* Serious problems with mobility.
* A history of neurological, mental, or substance abuse disorders.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participants will self-identify their gender orientation.
Enrollment: 402 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Increased physical activity | This effect should be observable (1) at the Week-4 post-test, (2) the Week-8 post-test, and (3) the 6-Month post-test.
  We expect that participants significantly increase their engagement in physical activity as assessed by an accelerometer.

CONTACTS AND LOCATIONS:
Overall Officials: Manfred K. Diehl, PhD, Principal Investigator — Colorado State University
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brothers A, Diehl M. Feasibility and Efficacy of the AgingPlus Program: Changing Views on Aging to Increase Physical Activity. J Aging Phys Act. 2017 Jul;25(3):402-411. doi: 10.1123/japa.2016-0039. Epub 2016 Dec 5. PMID 27918687
- [Background] Diehl M, Nehrkorn-Bailey A, Thompson K, Rodriguez D, Li K, Rebok GW, Roth DL, Chung SE, Bland C, Feltner S, Forsyth G, Hulett N, Klein B, Mars P, Martinez K, Mast S, Monasterio R, Moore K, Schoenberg H, Thomson E, Tseng HY. The AgingPLUS trial: Design of a randomized controlled trial to increase physical activity in middle-aged and older adults. Contemp Clin Trials. 2020 Sep;96:106105. doi: 10.1016/j.cct.2020.106105. Epub 2020 Aug 11. PMID 32791322
- [Background] Nehrkorn-Bailey AM, Rodriguez D, Forsyth G, Braun B, Burke K, Diehl M. Change in Views of Aging, Physical Activity, and Physical Health Over 8 Weeks: Results From a Randomized Study. J Aging Phys Act. 2023 Jan 28;31(4):666-678. doi: 10.1123/japa.2022-0133. Print 2023 Aug 1. PMID 36708712
- [Derived] Diehl M, Tseng HY, Rebok GW, Li K, Nehrkorn-Bailey AM, Rodriguez D, Chen D, Roth DL. Testing the purported mechanisms of the AgingPLUS intervention: Effects on physical activity outcomes. Psychol Aging. 2025 Jun;40(4):355-370. doi: 10.1037/pag0000893. Epub 2025 Apr 10. PMID 40208719
- [Derived] Tseng HY, Chasteen AL, Diehl M. Examining the malleability of implicit views of aging in middle-aged and older adults. Psychol Aging. 2025 Mar;40(2):147-158. doi: 10.1037/pag0000867. Epub 2024 Nov 25. PMID 39585776
- See also: Digital Object Identifier to the citation — https://doi.org/10.1123/japa.2016-0039

DOCUMENTS (1):
  • Informed Consent Form (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/48/NCT03299348/ICF_000.pdf